CLINICAL TRIAL: NCT03109158
Title: Phase I/II Clinical Trial of NC-6004 in Combination With 5-FU and Cetuximab as First-line Treatment in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: NC-6004 With 5-FU and Cetuximab for Treatment of Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NanoCarrier Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NC-6004-008
Record Dates: First submitted 2017-03-22; First posted 2017-04-12 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: squamous cell carcinoma; head; neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — demplatin pegraglumer; Cetuximab; Fluorouracil

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NC-6004 and 5-FU (Experimental): Phase I, continual reassessment method, dose-escalation study to determine the maximum tolerated dose (MTD) and an RPII dose of NC-6004 in patients with recurrent or metastatic squamous cell carcinoma of the head and neck.
  In Part 1, patients will be assigned to receive cetuximab followed by NC-6004 and 5-FU.
  Phase II, adaptive, open-label expansion study evaluating the activity, safety, and tolerability of NC-6004 in patients with recurrent or metastatic squamous cell carcinoma of the head and neck at the RPII dose identified in Part 1.
  In Part 2, all patients will receive NC-6004 at the RPII dose established in Part 1, in combination with cetuximab and 5-FU according to the same schedule as used in Part 1.
  Interventions: Drug: NC-6004; Drug: Cetuximab; Drug: 5-FU

INTERVENTIONS:
Drug: NC-6004 — NC-6004 provided by NanoCarrier
Drug: Cetuximab — Commercially Available
Drug: 5-FU — Commercially Available

SUMMARY:
Part 1 of this study will establish a recommended Phase II (RPII) dose for the triplet combination of NC-6004 plus 5-Fluorouracil (5-FU) and cetuximab. Part 2 will provide the efficacy signal of the triplet combination in this patient population.

DETAILED DESCRIPTION:
NC-6004 is a polymeric micelle-containing cisplatin as an active moiety. The nanoparticle provides sustained release of the active moiety and utilizes the enhanced permeability and retention effect to target release of platinum to tumors. Currently available nonclinical data and enhanced pharmacokinetics suggest that NC-6004 has the potential to be more active than cisplatin, with increased tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage III/IV recurrent and/or metastatic squamous cell carcinoma of the head and neck not suited for local therapy
* Measurable disease, as defined by RECIST v1.1
* ECOG performance status 0-1
* Adequate bone marrow reserve
* Adequate liver and renal function
* Have a negative pregnancy test result at Screening for females of childbearing potential
* Male patients must agree to use a condom during treatment and for 90 days after dosing and must agree not to donate sperm for 90 days after dosing
* Women of childbearing potential are willing to agree to use 1 of the study-defined effective methods of birth control from the time of study entry to 6 months after the last day of treatment
* Reasonably recovered from preceding major surgery as judged by the investigator or no major surgery within 4 weeks prior to the start of Day 1 treatment

Exclusion Criteria:

* Nasopharyngeal carcinoma
* Prior systemic chemotherapy, except if given as part of a multimodal treatment for locally advanced disease which was completed more than 3 months before Day 1 or more than 6 months prior to Day 1 if platinum-based
* Concomitant anticancer therapy, systemic immune therapy, or hormonal therapy as cancer therapy
* Unresolved toxicity from all radiation, adjuvant/ neoadjuvant chemotherapy, other targeted treatment including investigational treatment
* History of thrombocytopenia with complications
* Known hypersensitivity to platinum compounds
* Pregnant or breastfeeding
* Active infection (infection requiring intravenous antibiotics)
* Uncontrolled hypertension
* Malignancies other than head and neck cancer within 5 years prior to Day 1 of treatment, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* Signs or symptoms of organ failure, major chronic illnesses other than cancer, or any concomitant medical or social conditions which, in the opinion of the investigator, make it undesirable for the patient to participate in the study, or which could jeopardize compliance with the protocol
* Have experienced any of the following within the 6-month period prior to Screening: unstable angina pectoris, clinically significant coronary artery disease, cerebrovascular accident, transient ischemic attack, cardiac failure with known ejection fraction less than 40%, or cardiac arrhythmia
* Any investigational treatment within 30 days or 5 half-lives, whichever is longer, of Day 1 of treatment
* Patient is unwilling or unable to comply with study procedures, or is planning to take vacation for 7 or more consecutive days during the treatment phase of the study without prior consent from the medical monitor
* Any other medical or social condition that, in the opinion of the investigator, would not permit the patient to complete the study or sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
RPII dose for the combination of NC-6004 plus 5-FU plus cetuximab. | Up to day 90
  Part 1: To determine dose limiting toxicities and the RPII dose
Progression free survival in patients following treatment with NC-6004 plus 5-FU plus cetuximab. | Up to day 90
  Part 2: To determine the median PFS in patients with recurrent or metastatic squamous cell carcinoma of the head and neck after treatment with NC-6004 plus cetuximab plus 5-FU.

SECONDARY OUTCOMES:
Overall response rate | Up to day 90
  To evaluate overall response rate (ORR), duration of response (DOR), disease control rate (DCR = complete response [CR] + partial response [PR] +stable disease), duration of stable disease (DSD), and overall survival (OS).
EORTC QLQ-C30 | Up to day 90
  Least squares mean estimates for health-related quality of life (HRQOL) scores over time
QLQ-Head and Neck 35 | Up to day 90
  Least squares mean estimates for health-related quality of life (HRQOL) scores over time

OTHER OUTCOMES:
Incidence and severity of AEs and laboratory abnormalities | Up to day 90
  Incidence and severity of AEs and laboratory abnormalities, according to the NCI CTCAE v4.03 criteria.
Occurrence of SAEs and treatment discontinuations due to AEs | Up to day 90
  Adverse events will be summarized by dose level, in subsets of all TEAEs, and by all treatment-related AEs. Clinical laboratory and vital sign measurements will be summarized by dose level and change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Osada, Study Director, Study Director — NanoCarrier Co., Ltd.
Locations (20):
- United States (10):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Intermountain Precision Genomics, Billings, Montana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Bulgaria (2):
  - Complex Oncology Center - Shumen EOOD, Shumen
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
- Hungary (3):
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem, Pécs
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
- Romania (5):
  - Coltea Clinical Hospital, Bucharest
  - Prof Dr I Chiricuta Institute of Oncology, Cluj-Napoca
  - Oncology Center Sfantul Nectarie, Craiova
  - Euroclinic Oncology Center SRL, Iași
  - Institutul Regional de Oncologie Iasi, Iași